CLINICAL TRIAL: NCT03678909
Title: Cardiac Biomarkers in Patients With Single Ventricle Physiology
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Marc Anders, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-42776
Record Dates: First submitted 2018-09-16; First posted 2018-09-20 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Hypoplastic Left Heart; Congenital Heart Disease; Cyanotic Congenital Heart Disease; Cardiac Disease
Keywords: Troponin; BNP; Biomarkers; Hypoplastic Left Heart; Norwood; DKS
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Heart Defects, Congenital; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypoplastic Left Heart Disease: Patients with congenital hypoplastic left heart disease who will undergo surgical palliation with Norwood procedure or DKS or Damus-Kaye-Stansel procedure
  Interventions: Procedure: Norwood Palliation / DKS / Damus-Kaye-Stansel procedure

INTERVENTIONS:
Procedure: Norwood Palliation / DKS / Damus-Kaye-Stansel procedure — Norwood Palliation / DKS / Damus-Kaye-Stansel procedure

SUMMARY:
All neonates with congenital heart disease undergoing stage one palliation (Norwood procedure, Damus-Kaye-Stansel procedure) at Texas Children's Hospital will be regularly monitored for B-type natriuretic peptide (BNP) and Troponin level before the surgical procedure, on arrival to the cardiac intensive care unit after their surgical procedure, every 6 hours during the first 24 hours of the post-operative period, followed by daily levels for the first week, and then weekly during patient's regular laboratory work up schedule.

These cardiac biomarkers are linked to demographic, hemodynamic, respiratory, pharmacological data available via Sickbay.

DETAILED DESCRIPTION:
All neonates with congenital heart disease undergoing stage one palliation (Norwood procedure, Damus-Kaye-Stansel procedure) at Texas Children's Hospital will be regularly monitored for B-type natriuretic peptide (BNP) and Troponin level before the surgical procedure, on arrival to the cardiac intensive care unit after their surgical procedure, every 6 hours during the first 24 hours of the post-operative period, followed by daily levels for the first week, and then weekly during patient's regular laboratory work up schedule.

These cardiac biomarkers are linked to demographic, hemodynamic, respiratory, pharmacological data available via Sickbay.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Hypoplastic Left Heart Syndrome as congenital heart disease as a neonate

Exclusion Criteria:

Other diagnosis of congenital heart disease than Hypoplastic Left Heart Syndrome Patients older than 30 days

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonate with Hypoplastic Left Heart Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Mortality | 3- 6 months depending on second stage procedure
  Mortality up to anticipated Glenn Procedure

SECONDARY OUTCOMES:
NEC | 3- 6 months depending on second stage procedure
  Incidence of Necrotizing enterocolitis
Reintubation | 3- 6 months depending on second stage procedure
  Incidence of Reintubation
Cath intervention | 3- 6 months depending on second stage procedure
  Incidence of cath interventions

CONTACTS AND LOCATIONS:
Overall Officials: Marc M Anders, ND, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
The data is blinded to other study investigators.